CLINICAL TRIAL: NCT05353517
Title: Non-invasive Assessment of Brain and Spinal Synaptic Plasticity in Patients Affected by Movement Disorders
Brief Title: Non-invasive Assessment of Synaptic Plasticity
Acronym: NEUROPLAST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Antonio Suppa, Prof, MD, PhD, Neuromed IRCCS
Other Study IDs: NEUR_03
Record Dates: First submitted 2022-04-20; First posted 2022-04-29 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Movement Disorders; Parkinson Disease
MeSH Terms: conditions — Movement Disorders; Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Subjects: Device: focal muscle vibration to induce spinal plasticity theta burst stimulation and paired associative stimulation to induce plasticity in M1
  Interventions: Device: Device: focal muscle vibration and theta burst stimulation
- Patients with Parkinson's disease: Device: theta burst stimulation and paired associative stimulation to induce plasticity in M1 Device: focal muscle vibration to induce spinal plasticity
  Interventions: Device: Device: focal muscle vibration and theta burst stimulation

INTERVENTIONS:
Device: Device: focal muscle vibration and theta burst stimulation — non invasive techniques of neuromodulation for inducing plasticity in M1 and spinal cord

SUMMARY:
The pathophysiological mechanisms underlying Movement Disorders, including Parkinson's disease, have been related to altered synaptic plasticity affecting several structures of the central nervous system. Although several previous neurophysiologic investigations have shown abnormal long-term potentiation and depression-like plasticity in M1, other regions crucially involved in motor planning and execution, including the spinal cord, have been studied less. Parkinson's disease arises from the progressive loss of dendritic spines followed by atrophy of specific cortical (i.e. M1) and subcortical structures (i.e. putamen). These structural changes are responsible for the main clinical features of PD such as bradykinesia and rigidity. The present research project aims to probe non-invasively the main pathophysiologic mechanisms underlying altered synaptic plasticity in M1 and spinal cord and their relationship in a cohort of patients with movement disorders, including Parkinson's disease. More in detail, the investigators will use specific methodologies able to induce plasticity, including the repetitive transcranial magnetic stimulation (TMS), concerning the M1 and the focal muscle vibration, regarding the spinal cord. The neuromodulation protocol will imply 2 separate sessions, randomly scheduled to take into account the effect of the symptomatic pharmacologic treatment. Furthermore, patients will be randomly assigned to sham or real non-invasive stimulation groups. Before and after the stimulation protocol, the investigators will collect specific clinical as well as neurophysiologic measures (i.e., thresholds) according to standardized procedures. In conclusion, the goal of the study is to investigate the abnormal plasticity in the M1 and spinal cord in patients affected by specific movement disorders, through non-invasive techniques.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of Parkinson's disease

Exclusion Criteria:

* psychiatric disorders, including severe congnitive loss and depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 25 patients with PD 25 HS
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Analysis of neurophysiologic measures | baseline
  Rest motor threshold
Analysis of neurophysiologic measures | baseline
  Active motor threshold
Analysis of neurophysiologic measures | through study completion, an average of 1 year
  Amplitude of motor evoked potentials
Analysis of neurophysiologic measures | through study completion, an average of 1 year
  H reflex
Analysis of neurophysiologic measures | through study completion, an average of 1 year
  input-output curve

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Neuromed, Pozzilli, Italy

IPD SHARING:
Plan to Share IPD: Undecided